CLINICAL TRIAL: NCT07283796
Title: A Phase I Clinical Study to Evaluate the Safety, Efficacy, and PK/PD Characteristics of HSK47977 Tablets in Subjects With Relapsed or Refractory Non-Hodgkin's Lymphoma
Brief Title: A Study to Assess PK, Safety and Efficacy of HSK47977 Tablets in Subjects With Relapsed or Refractory Non-Hodgkin's Lymphoma
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Haisco Pharmaceutical Group Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HSK47977-101
Record Dates: First submitted 2025-12-02; First posted 2025-12-16 (Actual); Last update posted 2025-12-19 (Actual); Status verified 2025-12

CONDITIONS: NHL

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Phase Ia (Dose Escalation Part): HSK47977 (Experimental): Phase 1a (Dose Escalation Part): dose escalation of HSK47977 at various dose levels
  Interventions: Drug: HSK47977
- Phase Ia (Extension Part): HSK47977 (Experimental): Phase 1a (Part B): dose extention of HSK47977 at certain dose levels
  Interventions: Drug: HSK47977
- Phase Ib: HSK47977 (Experimental): Phase 1b: dose expansion for HSK47977 at dose of RP2D（Recommended Phase II Dose）
  Interventions: Drug: HSK47977

INTERVENTIONS:
Drug: HSK47977 — Taken orally once daily.

SUMMARY:
This is a Phase I Clinical Study to Evaluate the Safety, Efficacy, and PK/PD Characteristics of HSK47977 Tablets in Subjects with Relapsed or Refractory Non-Hodgkin's Lymphoma.This study includes a Phase Ia dose-escalation stage and a Phase Ib dose-expansion stage, and it is expected to take approximately 2 years.

ELIGIBILITY:
Inclusion Criteria:

1. Voluntarily sign the informed consent form.
2. Age ≥18 years, with no gender restriction.
3. Pathologically confirmed patients with relapsed/refractory Non-Hodgkin Lymphoma (rrNHL).
4. Eastern Cooperative Oncology Group (ECOG) performance status score of 0 to 2.
5. Expected survival >3 months.
6. Presence of measurable lesions.
7. Adequate organ function.
8. Agreement to undergo pathological tissue biopsy.
9. Subjects of childbearing potential must agree to comply with the contraceptive requirements of the study.
10. No pregnancy plans from screening until at least 3 months after the last dose of the study drug, and voluntary use of effective contraceptive measures.

Exclusion Criteria:

1. Concurrent presence of other severe, unstable diseases/conditions that, in the investigator's judgment, make participation in this study unsuitable.
2. History of or current severe cardiovascular disease.
3. Poorly controlled blood pressure during the screening period.
4. Laboratory abnormalities identified by the investigator that may pose a risk to the subject's safety.
5. Electrocardiogram abnormalities determined by the investigator as potentially posing a risk to the subject's safety.
6. History of allergies to the investigational drug or its excipients.
7. Inability to discontinue prohibited medications as specified in the protocol during the screening period and throughout the entire study duration.
8. Any other conditions that may increase subject risk or interfere with the trial results.
9. Any other situations where the investigator deems the subject unsuitable for participation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110 (Estimated)
Dates: Start 2025-08-28 (Actual); Primary Completion 2027-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Maximum tolerated dose (MTD) | Within first 28 days of treatment
  Highest dose level at which under 33% of patients in a cohort experience DLT（dose limiting toxicity）

CONTACTS AND LOCATIONS:
Locations (1):
- Chinese Academy of Medical Sciences Blood Diseases Hospital, Tianjin, China

IPD SHARING:
Plan to Share IPD: No